CLINICAL TRIAL: NCT07029022
Title: Monthly Trajectories of Mood Improvement Following a Workplace Mindfulness Programme: A Randomised Controlled Pilot Trial
Brief Title: Monthly Mood Improvement After Workplace Mindfulness
Acronym: MBI-WORK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shinyu Kise (Other)
Responsible Party: Sponsor-Investigator, Shinyu Kise, Principal Investigator , Institute for Tourism and Health, General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital.
Organization: General Incorporated Foundation Ryukyuseimeisaiseikai, Ryusei Hospital. (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-02
Record Dates: First submitted 2025-06-04; First posted 2025-06-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Mental Health Mood Disturbance Occupational Stress
Keywords: Mindfulness Workplace Intervention POMS2 Presenteeism Fatigue Pilot Study Randomized Controlled Trial Japan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention Group (Experimental): Participants in this arm received a workplace mindfulness-based intervention consisting of three 90-minute workshops spaced four weeks apart. The program included psychoeducation, guided stretching, and focused-attention meditation, supplemented by 10-minute daily self-practice and lifestyle guidance.
  Interventions: Behavioral: Mindfulness-Based Intervention (MBI)
- Wait-list Control Group (No Intervention): Participants in this arm did not receive any intervention during the three-month observation period. They were offered the same mindfulness-based program after the study was completed.

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention (MBI) — This intervention consisted of three 90-minute in-person workshops delivered monthly over a three-month period. Content included psychoeducation, guided stretching, and focused-attention meditation. Participants were also encouraged to practice mindfulness at home for 10 minutes daily and to follow lifestyle guidance on diet and physical activity.
  Arms: Mindfulness-Based Intervention Group

SUMMARY:
This randomized controlled pilot trial investigates the effects of a brief workplace mindfulness-based intervention (MBI) on mood among full-time employees in Japan. Twenty-five participants are randomly assigned to either the MBI group or a wait-list control group. The MBI group receives three 90-minute workshops spaced four weeks apart, along with daily home mindfulness practice. Mood is assessed monthly over three months using the Japanese version of the Profile of Mood States 2 (POMS2). The primary outcome is Total Mood Disturbance (TMD). This study is approved by the Ryusei Hospital Institutional Review Board and conducted as a feasibility trial.

DETAILED DESCRIPTION:
This pilot randomized controlled trial aims to evaluate the month-by-month effects of a low-intensity workplace mindfulness-based intervention (MBI) on mood among full-time employees in a healthcare setting in Okinawa, Japan. Participants are assigned in a 1:1 ratio to either the MBI group or a wait-list control group. The intervention consists of three 90-minute in-person workshops delivered at monthly intervals, incorporating psychoeducation, guided stretching, and focused-attention meditation. Participants in the MBI arm are also encouraged to practice mindfulness at home for 10 minutes per day. Mood is assessed at baseline and monthly over three months using the Japanese POMS2 Short Form. The primary endpoint is change in Total Mood Disturbance (TMD); secondary outcomes include fatigue (measured via a visual analogue scale) and presenteeism (measured via Single-Item Presenteeism Question, the University of Tokyo single-item edition (SPQ) ). Linear mixed-effects models are used for statistical analysis. The study is approved by the Ryusei Hospital Institutional Review Board (Approval No. 2024-02) and conducted as a feasibility study without prospective registration.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employment
* Age 20 years or older
* Provided written informed consent

Exclusion Criteria:

* Current or past psychiatric disorder
* Any medical condition deemed incompatible with study participation

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Change in Total Mood Disturbance (TMD) | Baseline to Month 3
  Total Mood Disturbance (TMD) score derived from the Japanese short form of the Profile of Mood States 2 (POMS2®). Monthly assessments were conducted over a three-month period. Higher scores indicate greater mood disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryusei Hospital, Naha, Okinawa, Japan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) underlying the primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and supporting documents will be available beginning 6 months after publication of the results and will remain available for 36 months.
Access Criteria: Qualified researchers with a methodologically sound proposal may request access to the data. Requests will be reviewed by the study team. A data use agreement will be required prior to data sharing.

REFERENCES:
- See also: Institute for Tourism and Health, Ryusei Hospital — https://www.ryusei.or.jp/checkup/Consulting#description-con-1